CLINICAL TRIAL: NCT02468440
Title: Evaluation of ESPAIR, an Educational Therapy's Program of Patients With Renal Insufficiency Before Kidney Transplant
Acronym: ESPAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14 7314 02; 2015/20 (Registry Identifier: CPP SOOM III)
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Renal Insufficiency
Keywords: renal insufficiency; kidney transplant; educational therapy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESPAIR (Experimental): Patients with an educational therapy's program since registration in transplant list.
  Interventions: Other: ESPAIR
- normal care (No Intervention): Patients without educational therapy

INTERVENTIONS:
Other: ESPAIR — ESPAIR is an educational therapy's program with 6 group session,and if patients ask for it, individual session are possible
  Arms: ESPAIR

SUMMARY:
Treatment care of end-stage renal insufficiency is an important public health issue. The balance between patients waiting for a kidney transplant and available graft raises questions. Because of the non-adherence, risk of graft loss is increased to 7 times so in this trial patients will experiment an educational therapy's program as soon as they register on the transplant list.

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal insufficiency on dialysis or not
* Registered on transplant list

Exclusion Criteria:

* Patient with psychological disorder
* transplantation from living donor
* Patients with renal transplant antecedent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Quality of life Questionnaire | 6 months
  Quality of life 6 months after registration on transplant list.

SECONDARY OUTCOMES:
Quality of life Questionnaire | One year
  Quality of life one year after registration on transplant list.
Quality of life Questionnaire | 1 day
  Quality of life on the day of the transplantation
Composite measure of impact of educational therapy's program | 6 months
  Impact of educational therapy's program on anxiety, knowledge to prepare transplant, life hygiene, and patient compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Laure Esposito, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Chu Toulouse, Toulouse, France